CLINICAL TRIAL: NCT06713044
Title: The Effect of Quranic Recitation and Classical Music on Postoperative Pain Intensity and Interleukin-6 Levels in Lower Limb Orthopedic Surgery with Intrathecal Anesthesia
Brief Title: Effect of Quranic Recitation and Classical Music on Pain Intensity and Interleukin-6 Levels After Lower Limb Orthopedic Surgery with Intrathecal Anesthesia
Acronym: QRCM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Jenderal Soedirman (Other)
Responsible Party: Principal Investigator, Guruh Perkasa, principal investigator, Universitas Jenderal Soedirman
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 420/08774
Record Dates: First submitted 2024-11-24; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Pain; Pain, Postoperative; Inflammation; Orthopedic Surgical Procedures
Keywords: Quranic Recitation; Classical Music Therapy; Pain Management; Inflammation IL 6; Non-Pharmacological Intervention
MeSH Terms: conditions — Pain; Pain, Postoperative; Inflammation; Agnosia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled trial with a parallel assignment study design. Participants will be randomly allocated to one of three groups:
  Murottal Group: Participants will listen to selected Islamic recitations (murottal) as a therapeutic intervention during their postoperative recovery.
  Classical Music Group: Participants will listen to selected classical music pieces to evaluate its impact on postoperative pain and inflammation.
  Standard Care Group: Participants will receive standard postoperative care without any additional therapeutic interventions.
  The goal is to assess and compare the effectiveness of murottal and classical music in reducing postoperative pain intensity and inflammation (measured by interleukin 6 levels), compared to the standard care. Randomization ensures unbiased distribution among the groups, and the parallel design enables simultaneous assessment of the interventions' effects in different groups.
Who Masked: Participant
Masking Description: participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Arm 1: Murottal Therapy (Experimental): Arm 1: Murottal Therapy
  Intervention: Participants in this group will listen to selected recitations of Islamic verses (murottal) as a non-pharmacological intervention during their postoperative recovery.
  Interventions: Device: Murottal Therapy Intervention Name: Murottal (Islamic verse recitation)
- Arm 2: Classical Music Therapy (Experimental): Intervention: Participants in this group will listen to selected classical music compositions during their recovery from lower extremity orthopedic surgery with spinal anesthesia.
  Interventions: Device: Classical Music Therapy Intervention Name: Classical Music Listening
- Arm 3: Standard Care (Experimental): Participants in this group will receive standard postoperative care following their surgery, without any additional interventions.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Device: Murottal Therapy Intervention Name: Murottal (Islamic verse recitation) — To evaluate whether murottal recitations can reduce postoperative pain intensity and lower interleukin 6 levels, which are indicative of inflammation.
  Arms: Arm 1: Murottal Therapy
Device: Classical Music Therapy Intervention Name: Classical Music Listening — To evaluate the impact of classical music on reducing postoperative pain intensity and interleukin 6 levels in the body, thereby managing inflammation.
  Arms: Arm 2: Classical Music Therapy
Other: Standard Care (in control arm) — To serve as a control group no intervention
  Arms: Arm 3: Standard Care

SUMMARY:
The goal of this study is to determine the effect of murottal and classical music on postoperative pain intensity and interleukin 6 levels in patients undergoing lower extremity orthopedic surgery with spinal anesthesia. This study also aims to evaluate whether these therapies can help reduce pain and influence the body's inflammatory response.

Main questions to be answered:

Can murottal or classical music reduce postoperative pain intensity in patients? Can the use of murottal or classical music lower the levels of interleukin 6, an inflammatory marker, in patients after lower extremity orthopedic surgery?

Participants will:

Listen to murottal or classical music during their lower extremity orthopedic surgery with spinal anesthesia.

Measure pain intensity and interleukin 6 levels before and after the intervention to assess the effect of the therapy.

Undergo routine checkups to ensure the safety and success of the therapy. This study aims to provide a deeper understanding of the use of non-pharmacological therapies such as murottal and classical music in managing pain and the inflammatory response in patients after orthopedic surgery.

DETAILED DESCRIPTION:
This study aims to explore the impact of murottal (recitations of Islamic verses) and classical music on postoperative pain intensity and interleukin 6 levels in patients undergoing lower extremity orthopedic surgery with spinal anesthesia. Murottal and classical music are considered non-pharmacological interventions and have been suggested to have a calming effect that may help reduce pain and manage inflammation.

During the study, participants will be randomly assigned to receive either murottal, classical music, or standard postoperative care. Participants in the murottal group will listen to selected recitations durante operation, while participants in the classical music group will listen to classical music compositions.

Pain intensity will be assessed using a numeric rating scale (NRS) both before and after the intervention. Interleukin 6 levels, an inflammatory marker, will be measured using blood samples taken at the same intervals.

The goal is to determine whether these therapeutic interventions can help reduce pain and inflammation, as indicated by interleukin 6 levels, compared to standard care alone. Regular check-ups will be conducted to monitor safety and ensure the success of the therapy.

The findings of this study will help provide insights into the potential use of non-pharmacological interventions, such as murottal and classical music, in managing pain and inflammation in postoperative patients, with the potential to improve recovery outcomes

ELIGIBILITY:
Inclusion Criteria:

1. All Muslim patients who are scheduled for elective lower extremity orthopedic surgery during the study period.
2. Patients aged 18 to 60 years.
3. Patients who agree to participate in the study.
4. Lower extremity orthopedic surgery (ORIF, OREF, and bone replacement) with a minimum surgery duration of 60 minutes.

Exclusion Criteria:

1. Patients with consciousness disorders
2. Patients with neurological disorders
3. Patients with cognitive disorders
4. Patients with more than 3 spinal attempts
5. Patients with hearing impairments
6. BMI < 18 and > 39 kg/m²

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Postoperatively | Timepoint: Pre-treatment (baseline, 10 minute before surgery) and post-treatment (30 minute post-surgery)
  Primary Outcome Measure 1: Pain Intensity Postoperatively Description: This measure will assess the intensity of pain experienced by participants after surgery.
  Method of Measurement: Numeric Rating Scale (NRS), where participants rate their pain on a scale from 0 (no pain) to 10 (worst pain imaginable).
Interleukin-6 (IL-6) Levels Postoperatively | Timepoint: Pre-treatment (baseline, 10 minute before surgery) and post-treatment (30 minute post-surgery)
  Primary Outcome Measure 2: Interleukin-6 Levels Postoperatively Description: This measure will evaluate the levels of IL-6, a marker for inflammation, following surgery.
  Method of Measurement: Blood sample analysis, expressed in picograms per milliliter (pg/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Margono Soekarjo Hospital, Purwokerto, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The Effect of Music Therapy on Pain, Anxiety and Vital Signs in Patients Undergoing Spinal Anaesthesia: A Randomized Controlled Trial Ibrahim Karagoz. et al.
- See also: The Effect of Perioperative Music on Medication Requirement and Hospital Length of Stay: A Meta-analysis — https://pubmed.ncbi.nlm.nih.gov/31356272/